CLINICAL TRIAL: NCT04167449
Title: Effects of Korean Red Ginseng Extract on Electrical Brain Activity in Elderly Subjects. A Prospective, Randomized, Double Blind, Placebo-controlled, 3-armed Cross-over Study
Brief Title: Effects of Korean Red Ginseng Extract on Electrical Brain Activity in Elderly Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EuroPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EP-1006
Record Dates: First submitted 2019-11-15; First posted 2019-11-18 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Brain Waves

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydroponic Red Ginseng (Active Comparator)
  Interventions: Dietary Supplement: HRG80 Hydroponic Red Ginseng
- Conventional White Ginseng (Active Comparator)
  Interventions: Dietary Supplement: Conventional White Ginseng
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: HRG80 Hydroponic Red Ginseng — Powdered root preparation of Panax ginseng standardized to 31.7 mg total ginsenosides
  Arms: Hydroponic Red Ginseng
Dietary Supplement: Conventional White Ginseng — Powdered root preparation of Panax ginseng standardized to 9.8 mg total ginsenosides
  Arms: Conventional White Ginseng
Dietary Supplement: Placebo — Visually identical placebo capsule containing rice flour
  Arms: Placebo

SUMMARY:
A prospective, randomized, double blind, placebo-controlled study to determine if a hydroponically-cultivated red ginseng preparation is superior to conventionally grown ginseng and placebo for positively affecting electrical activity of the brain during performance of various cognitive tasks.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be capable of giving informed consent.
* Acceptance of written consent to participate in the study after instruction in written and oral form (informed consent).

Exclusion Criteria:

* Subjects with acute or chronic diseases that are relevant to the study and asked for by the study staff are excluded:
* Acute or chronic disease with an impact on the study, which becomes obvious by case history or clinical examination.
* Clinically relevant allergic symptoms.
* Detection of alcohol at the time of initial examination (day SC) or on any study (positive alcohol test) or by case history.
* Consumption of clinically relevant medication during last 14 days before and during the active study period based on the notification of the subject or his case history.
* Consumption of medication with primarily central action (i.e. psychotropic drugs or centrally acting antihypertensive drugs). Known intolerance / hypersensitivity (allergy) to plant derived extracts or any of the ingredients of the investigational product (anamnestic).
* Consumption of unusual quantities or misuse of coffee (more than 4 cups a day), tea (more than 4 cups a day).
* Smoking in the study center on study days A, B, C and D.
* Participation in another clinical trial within the last 60 days.
* Bad compliance.
* Cancellation of informed consent.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Change in baseline electrical activity of the brain as measured by Quantitative Electroencephalogram for the hydroponic Korean red ginseng preparation versus conventional ginseng and placebo | Four weeks
  Responses of electric brain activity as spectral power in 17 different brain regions within 6 specially defined frequency ranges (delta, theta, alpha1, alpha2, beta1 and beta2) during cognitive performance: d2-test for attention (d2-Test).
Change in baseline electrical activity of the brain as measured by Quantitative Electroencephalogram for the hydroponic Korean red ginseng preparation versus conventional ginseng and placebo | Four weeks
  Responses of electric brain activity as spectral power in 17 different brain regions within 6 specially defined frequency ranges (delta, theta, alpha1, alpha2, beta1 and beta2) during cognitive performance: memory test (ME-Test).
Change in baseline electrical activity of the brain as measured by Quantitative Electroencephalogram for the hydroponic Korean red ginseng preparation versus conventional ginseng and placebo | Four weeks
  Responses of electric brain activity as spectral power in 17 different brain regions within 6 specially defined frequency ranges (delta, theta, alpha1, alpha2, beta1 and beta2) during cognitive performance: concentration-performance-test with financial reward (CPT-Test).

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Dimpfel, PhD, Principal Investigator — NeuroCode AG
Locations (1):
- Clinical Labors of NeuroCode AG, Wetzlar, Germany